CLINICAL TRIAL: NCT07123545
Title: Feasibility, Safety and Efficacy Study of Autologous Neoantigen-Specific T-Cell Therapy (iNeo-Vac-T01) in Advanced Hepatocellular Carcinoma Patients
Brief Title: Autologous Neoantigen-Specific T-Cell Therapy for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, Director physician, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZY-INEO-T01
Record Dates: First submitted 2025-07-30; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group（iNeo-Vac-P01+iNeo-Vac-T01） (Experimental): iNeo-Vac-P01 Personalized Neoantigen Peptide Vaccine Route of administration: Subcutaneous injection. Dosage: 0.3 mg per peptide. Administration schedule: Days 1, 4, 8, 15, 22, 52, and 82 (relative to treatment initiation).
  iNeo-Vac-T01 Personalized Cell Therapy (initiated at Week 9) Route of administration: Intravenous infusion. Dosing regimen: "3+3" dose escalation design. Dose Level 1: 5 × 10⁹ to 10 × 10⁹ cells. Dose Level 2: 1 × 10¹⁰ to 5 × 10¹⁰ cells.
  Lymphodepleting preconditioning regimen: Agents: Cyclophosphamide + Fludarabine. Timing: Administered prior to cell infusion.
  Post-infusion supportive therapy: Interleukin-2 (IL-2) support for 10 days.
  Interventions: Biological: iNeo-Vac-P01 Personalized Neoantigen Peptide Vaccine; Biological: iNeo-Vac-T01 Personalized T Cell Injection

INTERVENTIONS:
Biological: iNeo-Vac-P01 Personalized Neoantigen Peptide Vaccine — Administered subcutaneously at 0.3 mg/peptide on Days 1, 4, 8, 15, 22, 52, and 82, followed by booster immunizations every 2-3 months.
Biological: iNeo-Vac-T01 Personalized T Cell Injection — Administered via intravenous infusion: Dose Level 1: 5×10⁹ to 10×10⁹ cells; Dose Level 2: 1×10¹⁰ to 5×10¹⁰ cells.

SUMMARY:
The goal of this open-label, single-arm phase I/II clinical trial is to evaluate the feasibility, safety, and anti-tumor efficacy of the autologous neoantigen-specific T-cell therapy (iNeo-Vac-T01) in patients with advanced hepatocellular carcinoma who have failed second-line or later systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years (inclusive)
2. Histologically confirmed advanced hepatocellular carcinoma (HCC) with:

<!-- -->

1. Radiologically measurable disease per RECIST v1.1
2. Documented progression on ≥2 prior lines of systemic therapy 3.Life expectancy ≥6 months 4.ECOG performance status 0 or 1 5.Available archival or fresh tumor tissue sufficient for comprehensive genomic profiling OR existing whole-genome sequencing (WGS), whole-exome sequencing (WES), or RNA-sequencing data meeting prespecified quality thresholds 6.Adequate organ and marrow function:

(1)Hematologic:

1. White blood cell count (WBC) ≥3.0 × 10⁹/L
2. Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L
3. Hemoglobin ≥9.0 g/dL (≥5.6 mmol/L)
4. Platelet count ≥100 × 10⁹/L (2)Hepatic:

a.Total bilirubin ≤1.5 × upper limit of normal (ULN) (≤3 × ULN if liver metastases present) b.Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × ULN (≤5 × ULN if liver metastases present) (3)Renal:

1. Serum creatinine ≤1.5 × ULN OR
2. Calculated creatinine clearance (CrCl) ≥50 mL/min (Cockcroft-Gault formula) (4)Coagulation:

<!-- -->

1. International normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN AND activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless receiving therapeutic anticoagulation with stable INR/PT/aPTT within target range) 7.Reproductive Status:

   1. Women of childbearing potential (WOCBP): Negative serum pregnancy test within 7 days prior to treatment initiation AND agreement to use highly effective contraception during study participation and for ≥120 days after last study intervention
   2. Men: Agreement to use barrier contraception during study participation and for ≥120 days after last study intervention 8.Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

   Exclusion Criteria:

   1.History of other active malignancies within the past 5 years, except:
   1. Adequately treated basal cell or squamous cell skin cancer
   2. Carcinoma in situ of the cervix
   3. Other malignancies considered cured with minimal risk of recurrence (e.g., localized thyroid cancer) 2.Failure to identify therapeutically targetable neoantigens via genomic analysis 3.Prior allogeneic bone marrow, solid organ, or hematopoietic stem cell transplantation 4.Active or symptomatic central nervous system (CNS) metastases except:

   (1)Previously treated CNS metastases that are radiologically stable (no evidence of progression) for ≥4 weeks and (2)Asymptomatic and off corticosteroid/anticonvulsant therapy for ≥4 weeks prior to enrollment (3)Note: Leptomeningeal disease is excluded regardless of stability or treatment status.

   5.Active bacterial, fungal, or mycobacterial infection requiring systemic therapy (including untreated latent tuberculosis) 6.Active viral infections meeting any of the following:
   1. Detectable HBV DNA (if HBsAg positive or HBcAb positive)
   2. Detectable HCV RNA
   3. HIV infection (serologically confirmed)
   4. Active syphilis infection (serologically confirmed) 7.Active autoimmune disease requiring systemic immunosuppressive therapy (>10 mg prednisone equivalent daily) within the past 2 years, except:

   <!-- -->

   1. Vitiligo
   2. Type 1 diabetes mellitus
   3. Hypothyroidism stable on hormone replacement
   4. Psoriasis not requiring systemic therapy 8.Systemic immunosuppressive therapy (>10 mg prednisone equivalent per day) within 14 days prior to planned cell infusion (topical, inhaled, or ophthalmic corticosteroids are permitted) 9.Uncontrolled intercurrent illness including, but not limited to:

   (1)New York Heart Association (NYHA) Class III or IV congestive heart failure (2)Unstable angina pectoris (3)Uncontrolled cardiac arrhythmia (4)Uncontrolled hypertension (≥160/100 mmHg despite medication) (5)Clinically significant pulmonary disease 10.History of substance abuse or psychiatric/social condition that would impair ability to provide informed consent or comply with study requirements 11.History of severe (Grade ≥3) hypersensitivity reactions to vaccine components or investigational products, or any condition deemed by the investigator to pose an unacceptable risk for immunotherapy 12.Any condition that, in the opinion of the Investigator, would compromise patient safety or interfere with study participation or interpretation of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Successful Administration Rate of iNeo-Vac-T01 | Up to 3 years
  Proportion of enrolled patients who received the complete planned iNeo-Vac-T01 cell infusion.
Incidence of Adverse Events (AEs) | Up to 3 years
  Incidence of adverse events (AEs) graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, including serious adverse events (SAEs) .

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 3 years
  Defined as the time from the first administration of iNeo-Vac-P01 to the first documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause (whichever occurs first), or the time from the first administration of iNeo-Vac-T01 to the first documented disease progression per RECIST v1.1 or death from any cause (whichever occurs first). Disease progression is determined by investigator assessment of serial tumor imaging [Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)].
Objective Response Rate (ORR) | up to 3 years
  Defined as the proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 criteria.Disease progression is determined by investigator assessment of serial tumor imaging [Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)].
Neoantigen-Specific T Cell Response in Peripheral Blood | up to 3 years
  Vaccine-induced neoantigen-specific CD4⁺ and CD8⁺ T lymphocyte responses detected in peripheral blood using enzyme-linked immunospot (ELISpot) assay .

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No